CLINICAL TRIAL: NCT00308399
Title: A Double Blind, Randomized, Placebo-controlled, Single Center, Parallel Group Study to Evaluate the Effects of Itopride (100 mg and 200 mg t.i.d.) on Gastric Motor and Sensory Functions in Healthy Volunteers.
Brief Title: A Study to Evaluate the Effect of a Medicine on Gastric Functions in Healthy Volunteers.
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Axcan Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1099-05
Record Dates: First submitted 2006-03-27; First posted 2006-03-29 (Estimated); Last update posted 2011-03-23 (Estimated); Status verified 2011-03

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — itopride

INTERVENTIONS:
Drug: Itopride

SUMMARY:
A 7 day study which involves 2 nutrient drink tests, an ECG, a Scintigraphy scan, and a Sect scan. This study requires the participant to make 4 visits to the GCRC in the Charlton building but no overnight stays.

DETAILED DESCRIPTION:
A screening interview and symptoms assessment by the Bowel Disease Questionnaire (BDQ) and consent will be obtained prior to the studies at the testing facility (General Clinical Research Center, 7th floor, Charlton Building, Mayo Clinic). Smoking status will be recorded. Vitals and an electrocardiogram will be obtained. Following an initial screening, subjects will be randomized to itopride or identical placebo.

Day 1: The participant will report in a fasting condition (10 hours) to the study center early in the morning. All participants will undergo the nutrient drink test to assess maximum tolerated volume and postprandial symptoms PRIOR to ingesting any medication.

Day 2-7: The patients will take the study medication as prescribed that is a tablet 30 minutes before meals, three times per day. On days 6, 7 and 8, the morning and midday dose of the medication intake will occur in the clinical research center under supervision of the study staff.

Day 6: The participant will return fasting for 10 hours to the study center early in the morning. Scintigraphic gastric and small bowel transit measurement will be performed, with medication ingested at standard times (30 min prior to meal), and the 99mTc-sulfur colloid labeled egg meal ingested 30 minutes after the morning dose of study medication. Imaging will be taken for 6 hours. Vitals and an electrocardiogram will be obtained Day 7: All participants will undergo a repeat nutrient drink test to assess postprandial symptoms at maximal satiety and 30 minutes after drug ingestion. The satiety study will be completed once a maximum tolerated volume is achieved, and the 30 minute post-meal questionnaire will be completed.

Day 8: The participant will return fasting to the study center early in the morning. Participants will undergo SPECT imaging to evaluate fasting gastric volume starting 30 minutes after ingestion of study medication. The participant will then ingest 300 ml of the nutrient drink Ensure", and postprandial gastric volumes will be calculated as described previously (41-46). Vitals will be obtained.

ELIGIBILITY:
1. Non-pregnant, non-breastfeeding females;
2. 18- 45 years old
3. Body mass index between 20 and 32 kg/m2
4. No alarm indicators on clinical assessment (weight loss of more than 7kg, bleeding, recent recurrent vomiting, progressive dysphagia).
5. No history suggestive of small bowel obstruction

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2005-11; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Post-prandial post drug volume-fasting post drug volume (gastric accommodation).

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas J. Talley, M.D., Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States